CLINICAL TRIAL: NCT05269056
Title: Early Detection of Stage I-II Gastric Cancer Using Plasma Cell-free DNA Fragmentomics
Brief Title: Early Detection of Gastric Cancer Using Plasma Cell-free DNA Fragmentomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Nanjing Geneseeq Technology Inc. (Industry)
Responsible Party: Principal Investigator, Xiangdong Cheng, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2021-295
Record Dates: First submitted 2022-02-28; First posted 2022-03-07 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Early Gastric Cancer
Keywords: Gastric cancer; Early stage; Plasma Cell-free DNA; Fragmentomic assay
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Cell-free DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage I-II gastric cancer: Cell-free DNA collected from plasma samples of 200 patients with stage I-II gastric cancer will undergo whole-genome sequencing
- Healthy controls: Cell-free DNA collected from plasma samples of 100 non-cancer individuals will serve as controls

SUMMARY:
The purpose of this study is to enable non-invasive early detection of gastric cancer in high-risk populations through the establishment of a multimodal machine learning model using plasma cell-free DNA fragmentomics. Plasma cell-free DNA from early stage gastric cancer patients and healthy individuals will be subjected to whole-genome sequencing. Features, such as cell-free DNA fragmentation, copy number variations and microbiome, will be assessed to generate this model.

DETAILED DESCRIPTION:
Improvement in the specificity of early cancer detection reduces financial and mental burdens from unnecessary screenings. Advances in liquid biopsy approaches have expanded the clinical scope of cell-free DNA analysis in cancer early detection, by moving away from cell-free DNA methylome toward an integrative approach that enables the simultaneous assessment of multimodal cell-free DNA features. Integration of liquid biopsy-based cancer early detection into the clinic requires optimization of detection techniques, large-scale studies and prospective clinical validation. In the early detection of gastric cancer, the top research priorities are to identify relevant target features and to improve the sensitivity and specificity of detection. This large-scale early detection study will randomly enroll 200 stage I/II pathologically diagnosed gastric patients and 100 age- and sex-matched healthy individuals upon providing written informed consent. Plasma samples will be collected and extracted cell-free DNA will be subjected to whole genome sequencing. We aimed to incorporate genome-wide copy number variations, cell-free DNA fragmentomics, and microbiome features into the development of a multimodal biomarker-based prediction model.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum 18 years
* Participants must have histologically and/or cytologically confirmed stage I/II gastric cancer
* Full access to the patients' clinical and pathological records
* Ability to understand and the willingness to sign a written informed consent document
* Non-cancer controls are sex- and age-matched individuals without presence of any tumors or nodules or any other severe chronic diseases through systematic screening

Exclusion Criteria:

* Participants must not be pregnant or breastfeeding
* Participants must not have prior cancer histories or a second non-gastric malignancy
* Participants must not have had any form of cancer treatment before enrollment or plasma collection, including surgery, chemotherapy, radiotherapy, targeted therapy and immunotherapy
* Participants must not present medical conditions of fever or have acute or immunological diseases that required treatment 14 days before plasma collection
* Participants who underwent organ transplant or allogenic bone marrow or hematopoietic stem cell transplantation
* Participants with clinically important abnormalities or conditions unsuitable for blood collection
* Any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction, major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or psychiatric illness/social situations that would limit compliance with study requirements or influence patient signing the written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 200 stage I/II gastric cancer patients and 100 non-cancer controls
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve of the model for detecting stage I/II gastric cancer | 2 years
  The area under curve of the model for the ultrasensitive early detection of stage I/II gastric cancer would be evaluate

SECONDARY OUTCOMES:
Sensitivity of the early detection model | 2 years
  The sensitivity of the model for the ultrasensitive early detection of stage I/II gastric cancer would be evaluate
Specificity of the early detection model | 2 years
  The specificity of the model for the ultrasensitive early detection of stage I/II gastric cancer would be evaluate
Area under curve of the early detection model at sequencing depth downsampling | 2 years
  The area under curve of the model at sequencing depth downsampling for the ultrasensitive early detection of stage I/II gastric cancer would be evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, PhD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital；Cancer hospital of the university of chinese academy of sciences, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu P, Chen P, Wu M, Ding G, Bao H, Du Y, Xu Z, Yang L, Fang J, Huang X, Lai Q, Wei J, Yan J, Yang S, He P, Wu X, Shao Y, Su D, Cheng X. Multi-dimensional cell-free DNA-based liquid biopsy for sensitive early detection of gastric cancer. Genome Med. 2024 Jun 7;16(1):79. doi: 10.1186/s13073-024-01352-1. PMID 38849905